CLINICAL TRIAL: NCT00785954
Title: Inhibition of Delta-protein Kinase C for the Reduction of Infarct Size in Acute Myocardial Infarction
Brief Title: Safety and Efficacy Study of KAI-9803 to Treat Subjects With ST Elevation Myocardial Infarction [Heart Attack]
Acronym: PROTECTION AMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Collaborators: Bristol-Myers Squibb (Industry); The Cleveland Clinic (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KAI-9803-004; EudraCT: 2008-005140-16
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Myocardial Infarction; Cardiovascular Diseases; Pathologic Processes
Keywords: Heart Diseases; Myocardial Ischemia; Infarction; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases; Pathologic Processes; Heart Diseases; Myocardial Ischemia; Infarction | interventions — KAI 9803

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1: KAI-9803 (Experimental)
  Interventions: Drug: KAI-9803
- A2: KAI-9803 (Experimental)
  Interventions: Drug: KAI-9803
- A3: KAI-9803 (Experimental)
  Interventions: Drug: KAI-9803
- A4: Placebo (Placebo Comparator)
  Interventions: Drug: KAI-9803

INTERVENTIONS:
Drug: KAI-9803 — STEMI Subjects will be randomly assigned to receive either KAI-9803 or Placebo

SUMMARY:
The purpose of this study is to determine whether KAI-9803 is safe and effective in reducing infarct size in subjects with ST elevation myocardial infarction (heart attack) undergoing a percutaneous coronary intervention (PCI). A select number of sites will also participate in a substudy where eligible patients will undergo an additional procedure;cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Acute STEMI and has a planned emergent primary PCI procedure
* Continuous symptoms of cardiac ischemia and present to the primary PCI facility within 6 hours of symptom onset

Exclusion Criteria:

* Persistent systolic blood pressure < 90 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The effect of KAI-9803 on infarct size as assessed by CK-MB AUC | During the index hospitalization

SECONDARY OUTCOMES:
The effect of KAI-9803 on the incidence of the composite of cardiovascular death, heart failure, or serious ventricular arrhythmias | Within the first 3 months after Myocardial Infarction
The safety and tolerability of KAI-9803 by IV infusion to acute STEMI | Within the first 3 months after Myocardial Infarction
Assess left ventricular function by imaging | Within the first 3 months after Myocardial Infarction

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bell, MD, Study Director — KAI Pharmaceuticals, Inc; A.Michael Lincoff, MD, Principal Investigator — The Cleveland Clinic
Locations (126):
- United States (17):
  - Huntsville, Alabama
  - Escondido, California
  - Torrance, California
  - Tampa, Florida
  - Atlanta, Georgia
  - Downers Grove, Illinois
  - Lombard, Illinois
  - Peoria, Illinois
  - Valparaiso, Indiana
  - Omaha, Nebraska
  - Williamsville, New York
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Beaver, Pennsylvania
  - Danville, Pennsylvania
- Australia (11):
  - Bedford Park
  - Boxhill
  - Epping
  - Fremantle
  - Hobart
  - Kogarah
  - Liverpool
  - Parkville
  - Perth
  - St Leonards
  - Victoria
- Belgium (5):
  - Antwerp
  - Bonheiden
  - Brussels
  - Liège
  - Roeselare
- Canada (10):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Kitchner, Ontario
  - Newmarket, Ontario
  - Toronta, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - New Brunswick
- Czechia (10):
  - Brno
  - Hradec Králové
  - Karlovy Vary
  - Labem
  - Liberec
  - Olomouc
  - Ostrava
  - Pilsen
  - Prague
  - Zlín
- Denmark (4):
  - Aalborg
  - Copenhagen
  - Hellerup
  - Odense
- Finland (2):
  - Helsinki
  - Turku
- Germany (9):
  - Berlin
  - Halle
  - Hamburg
  - Heidelberg
  - Lübeck
  - Magdeburg
  - Mannheim
  - München
  - Rostock
- Hungary (5):
  - Budapest
  - Pécs
  - Szeged
  - Székesfehérvár
  - Zalaegerszeg
- Israel (9):
  - Afula
  - Ashkelon
  - BeerSheva
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Safed
  - Ẕerifin
- Italy (3):
  - Pesaro
  - Rome
  - Rozzano
- Netherlands (4):
  - Amsterdam
  - Nieuwegein
  - Rotterdam
  - Zwolle
- New Zealand (5):
  - Auckland
  - Christchurch
  - Dunedin
  - Hamilton
  - Nelson
- Norway (2):
  - Arendal
  - Bergen
- Poland (11):
  - Bialystok
  - Bielsko-Biala
  - Dąbrowa Górnicza
  - Gdansk
  - Gdynia
  - Krakow
  - Lubin
  - Poznan
  - Szczecin
  - Torun
  - Warsaw
- Portugal (3):
  - Almada
  - Amadora
  - Carnaxide
- Spain (8):
  - Alicante
  - Barcelona
  - El Palmar Murcia
  - León
  - Madrid
  - Santa Cruz de Tenerife
  - Seville
  - Vigo Pontevedra
- Sweden (8):
  - Gothenburg
  - Helsingborg
  - Linköping
  - Lund
  - Malmo
  - Örebro
  - Stockholm
  - Sundsvall

REFERENCES:
- [Derived] Lincoff AM, Roe M, Aylward P, Galla J, Rynkiewicz A, Guetta V, Zelizko M, Kleiman N, White H, McErlean E, Erlinge D, Laine M, Dos Santos Ferreira JM, Goodman S, Mehta S, Atar D, Suryapranata H, Jensen SE, Forster T, Fernandez-Ortiz A, Schoors D, Radke P, Belli G, Brennan D, Bell G, Krucoff M; PROTECTION AMI Investigators. Inhibition of delta-protein kinase C by delcasertib as an adjunct to primary percutaneous coronary intervention for acute anterior ST-segment elevation myocardial infarction: results of the PROTECTION AMI Randomized Controlled Trial. Eur Heart J. 2014 Oct 1;35(37):2516-23. doi: 10.1093/eurheartj/ehu177. Epub 2014 May 5. PMID 24796339